CLINICAL TRIAL: NCT07257081
Title: Effect of Combining Filling of the Posterior Superior Notch of the Humerus With a Coracoid Stop on the Rate of Return to Sports at the Same Level: a Randomized Study
Brief Title: Effect of Combining a Posterosuperior Humeral Notch Filling With a Coracoid Bone Block on the Rate of Return to Sport
Acronym: BUTEE2024
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-A02276-41
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic coracoid process resection (No Intervention): Arthroscopic coracoid process resection
- Arthroscopic coracoid process resection + filling of the posterosuperior notch of the humerus (Experimental): Arthroscopic coracoid process resection with filling of the posterosuperior notch of the humerus
  Interventions: Procedure: Filling of the posterior superior notch of the humerus

INTERVENTIONS:
Procedure: Filling of the posterior superior notch of the humerus — The intervention involves bringing part of the coracoid bone with the tendon attached to it onto the front of the glenoid cavity. The stop is secured with an endobutton. The additional procedure used in this study is filling the posterosuperior notch of the humerus. The filling technique involves placing two anchors, which causes tenodesis of the infraspinatus in the posterosuperior notch of the humerus.
  Arms: Arthroscopic coracoid process resection + filling of the posterosuperior notch of the humerus

SUMMARY:
The goal of this interventional study is to demonstrate the benefit of combining filling of the posterosuperior notch of the humerus with a coracoid stop on the rate of return to sports at the same level as before at 12 months post-surgery.

The level of sport will be categorized as recreational, competitive, or professional.

This is a prospective, single-center, comparative study of two parallel randomized groups, using a single-blind design.

The patients included will be randomized into two groups with a 1:1 ratio: one group will undergo the filling technique, while the second group will not. The rest of the surgery will be similar.

Randomization will be stratified according to initial athletic level.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient affiliated with or entitled to social security coverage
* Patient who has received informed consent about the study and signed a consent form
* Patient presenting with previous shoulder instability associated with a compromising humeral lesion determined by CT scan measurement

Exclusion Criteria:

* Patient non-compliant with follow-up over 1 year
* Recurrence of a previously operated shoulder
* Patient under judicial protection, guardianship, or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants returning to sports at the same level after surgery, in each arms, at 12months | 12 months
  Difference between the two arms for returning to sports at the same level as before, categorized into three levels: recreational, competitive, or professional, 12 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique St Jean Sud de France, Saint-Jean-de-Védas, France